CLINICAL TRIAL: NCT03425565
Title: A Phase II Study of Pembrolizumab in Patients With Advanced Gynaecological Clear Cell Cancer
Brief Title: A Study of Pembrolizumab in Patients With Advanced Gynaecological Clear Cell Cancer
Acronym: PEACOCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/17/0672
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-11

CONDITIONS: Clear Cell Tumor; Gynecologic Cancer; Advanced Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 3 weekly cycles of Pembrolizumab administered by IV

SUMMARY:
PEACOCC is a multi-centre, single arm, single stage phase II trial. The overall aim is to determine whether treatment with pembrolizumab is effective in patients with advanced clear cell gynaecological cancer.

ELIGIBILITY:
Main Inclusion Criteria:

1. Histological diagnosis of advanced clear cell ovarian (including primary peritoneal and fallopian tube), endometrial, vaginal, vulval or cervical cancer.
2. Have measurable disease based on RECIST 1.1.
3. Evidence of radiological disease progression.
4. Patient is willing to provide tissue from a newly obtained core or excisional biopsy of a tumour lesion at baseline, 6-8 weeks after start of treatment and at the time of progression.
5. ECOG Performance Status 0 or 1.
6. Patient has a life expectancy of at least 3 months from consent.
7. Received ≥ 1 line of prior chemotherapy .

Main Exclusion Criteria:

1. Has a known diagnosis of immunodeficiency or is receiving systemic steroid therapy at doses > 10mg prednisolone daily or equivalent or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
2. Has a known history of active TB (Bacillus Tuberculosis), Hepatitis B (e.g., HBsAg reactive), Hepatitis C or a known history of Human Immunodeficiency Virus (HIV).
3. Has symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis.
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids (at a dose >10mg predisolone daily or equivalent) or immunosuppressive drugs).
5. Has known history or evidence of active, non-infectious pneumonitis.
6. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
7. Has received a live vaccine within 30 days prior to the planned start of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Western General Hospital, Edinburgh
  - University College Hospital, London
  - The Christie Hospital, Manchester
  - Mount Vernon Hospital, Northwood
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kristeleit R, Devlin MJ, Clamp A, Gourley C, Roux R, Hall M, Nirsimloo R, Kounnis V, Sage L, Narayanan P, Herrington CS, Arora R, Farrelly L, Hughes L, Counsell N, Miller RE. Pembrolizumab in Patients With Advanced Clear Cell Gynecological Cancer: A Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2025 Apr 1;11(4):377-385. doi: 10.1001/jamaoncol.2024.6797. PMID 39913118